CLINICAL TRIAL: NCT07048028
Title: Evaluation of the Antibacterial Efficacy of Chitosan as an Irrigation Solution: A Randomized Controlled Clinical Trial
Brief Title: Chitosan Irrigation in Premolar Root Canal Therapy (Randomized Trial)
Acronym: CHITO-PRE RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ESRA DAĞCI (Other)
Responsible Party: Sponsor-Investigator, ESRA DAĞCI, Research Assistant Esra Dagci, Ordu University
Organization: Ordu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025000117-1
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Apical Periodontitis; Dental Pulp Necrosis; Root Canal Infection
MeSH Terms: conditions — Periapical Periodontitis; Dental Pulp Necrosis | interventions — Sodium Hypochlorite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chitosan irrigation (Experimental): Root canal irrigated with 0.2 % chitosan.
  Interventions: Drug: Chitosan Low Molecular Weight (20-200 Mpa.S)
- NaOCl and Chitosan irrigation (Experimental): Root canal irrigated with 10 mL of 2.5 % sodium hypochlorite (60 s contact), followed by 10 mL of 0.2 % chitosan solution (60 s contact). Final flush with 5 mL sterile saline
  Interventions: Drug: Chitosan Low Molecular Weight (20-200 Mpa.S); Drug: Sodium Hypochlorite
- NaOCl and EDTA irrigation (Experimental): Root canal irrigated with 10 mL of 2.5 % sodium hypochlorite (60 s contact), followed by 10 mL of 17 % EDTA solution (60 s contact). Final flush with 5 mL sterile saline.
  Interventions: Drug: Sodium Hypochlorite; Drug: EDTA chelating agents

INTERVENTIONS:
Drug: Chitosan Low Molecular Weight (20-200 Mpa.S) — A 0.2 % (w/v) low-molecular-weight chitosan solution (50-190 kDa, ≥75 % deacetylation) prepared fresh in 1 % acetic acid, pH ≈ 6.0. Ten mL is delivered into the root canal over 30 s and left in situ for an additional 30 s (total contact 60 s), followed by a 5 mL sterile saline flush
  Arms: Chitosan irrigation; NaOCl and Chitosan irrigation
Drug: Sodium Hypochlorite — Commercial 2.5 % (w/v) sodium hypochlorite endodontic irrigant. Ten mL is delivered over 30 s and left for 30 s (total contact 60 s), then flushed with 5 mL sterile saline
  Arms: NaOCl and Chitosan irrigation; NaOCl and EDTA irrigation
Drug: EDTA chelating agents — Ready-to-use 17 % EDTA solution (pH ≈ 7.3) for smear-layer removal. Ten mL is delivered over 30 s and left for 30 s (total contact 60 s), then flushed with 5 mL sterile saline
  Arms: NaOCl and EDTA irrigation

SUMMARY:
The goal of this clinical trial is to learn which of three common root-canal rinsing (irrigation) methods removes bacteria most effectively in adult patients who need root-canal treatment. The main questions it will answer are:

How much does a chitosan solution used alone lower the number of bacteria inside the root canal? Do the combinations sodium hypochlorite + chitosan or sodium hypochlorite + EDTA lower bacteria even more than chitosan alone? Researchers will compare the three irrigation methods to see which one achieves the greatest bacterial reduction.

What participants will do

Be randomly assigned to one of three groups:

Group 1: Chitosan only Group 2: Sodium hypochlorite followed by chitosan Group 3: Sodium hypochlorite followed by EDTA

Attend two clinic visits:

Visit 1:

Receive standard root-canal treatment under local anesthesia. Provide tiny paper-point samples from inside the canal before and after the assigned rinse (painless; takes seconds).

Visit 2 (about 1 week later):

Return for a check-up and final filling of the tooth. Record any pain or discomfort for the first three days after treatment in a simple diary (or by phone).

About 90 adults will take part. All procedures are routine in dental care, and there is no cost to participate. Participants may withdraw at any time and can ask the study dentist any questions throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agreed to participate in the study
* Systemically healthy patient
* Mandibular premolar teeth
* Teeth that respond negatively to thermal tests and EPT
* Patients who have not used antibiotics for at least 2 weeks

Exclusion Criteria:

* Teeth with previous primary root-canal treatment
* Pregnant patients
* Severely curved roots (>25° curvature)
* Canals with instrument separation during preparation
* Calcified (obliterated) canals

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-11-17 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Change in Intracanal Bacterial Load | Baseline (pre-instrumentation) to Immediate Post-instrumentation (sample processed ≤ 48 h)"
  Change in Intracanal Bacterial Load (log10 CFU/mL) From Baseline to Immediate Post-instrumentation

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Cakici, DDS, PhD, Principal Investigator — Ordu University Faculty of Dentistry
Locations (1):
- Ordu University, Ordu, Altınordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level log10 CFU/mL data (baseline and immediate post-instrumentation) will be available 12 months after publication. Researchers may request the dataset by emailing the Principal Investigator; a data-sharing agreement will be required.
Supporting Information: Study Protocol
Time Frame: Beginning 12 months after primary publication and ending 5 years after publication
Access Criteria: Access to the de-identified participant-level log10 CFU/mL dataset (baseline and immediate post-instrumentation) will be granted to qualified, non-commercial academic investigators.
  Requests must include a brief research proposal and proof of institutional ethics approval, and should be e-mailed to the Principal Investigator (dagci.esra.496@gmail.com). After approval and signature of a data-sharing agreement that prohibits re-identification or further redistribution, the dataset and data dictionary will be transferred via a secure, password-protected file-sharing service.
  No clinical charts, radiographs, consent forms, or ethics-committee documents will be shared. Data will be available beginning 12 months after primary publication, with no end date.